CLINICAL TRIAL: NCT02956824
Title: Incidence of Sacro-Iliac Joint Anomalies on MRI in Women Aged From 18 to 50 Years Old
Brief Title: Incidence of MRI Sacro-Iliac Joint Anomalies in Young Women
Acronym: MISIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9626
Record Dates: First submitted 2016-08-01; First posted 2016-11-07 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Women (Between 18 to 50 Years Old); Sacro-iliac Joints; Inflammatory Lesions; Structural Lesions; Axial Spondyloarthritis
Keywords: Magnetic Resonance Imaging (MRI); Sacro-iliac joints; Pelvis; Erosion; Fat deposit; Subchondral sclerosis; Bone marrow edema; Axial spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Standard care — Current care

SUMMARY:
Prospective multicenter study assessing the incidence of inflammatory and structural lesions seen on MRI of the SI joints in a consecutive population of women aged 18-50 years old.

The study hypothesis is SpA may be misdiagnosed on MRI in post partum women due to increased stress on the joint following pregnancy and childbirth, as MRI of the SI joints may show lesions that could mimics axial spondyloarthritis. The primary objective of this study is to determine the incidence of SI lesions seen at MRI in women. The secondary objectives are to compare the incidence and pattern of MRI inflammatory and structural lesions of the SI joints and to determine the factors associated with inflammatory or structural changes of the SI joints in a population of women. the investigators will especially compare the population of women within a year after childbirth versus the population of women who never gave birth or who gave birth over 24 months ago or more.

DETAILED DESCRIPTION:
500 women aged of 18 to 50 years old, including 100 women who gave birth within the year, referred to the Imaging department for pelvic MRI for the exploration of pelvic or gynecologic pathology will be recruited consecutively.

MRI will be performed on a 1.5 T MRI according to standardized exploration of the pelvis and will include axial T1-weighted sequences and T2STIR (or T2 fat sat or T2 Dixon) of maximum 6 mm thickness .

An additional Axial STIR sequence may be added as part of the research (duration 3 minutes), if the standard protocol does not include any STIR, T2 fat sat T2 or T2 Dixon sequence.

SI lesions will be assessed in a centralized randomized and independent review of all MR images by 2 musculoskeletal radiologists according to ASAS criteria.

Patients will complete a standardized questionnaire on the day of MRI to collect the following data : patient's and family history of chronic inflammatory disease, number and date of pregnancies, practice of sports, back pain, joint pain.

ELIGIBILITY:
Inclusion criteria:

* Women aged 18 to 50 years old
* MRI of the pelvis requested as part of an exploration of a gynecological or pelvic pathology
* Women who delivered within the year OR women who never gave birth or gave birth 24 months ago and over

Exclusion criteria:

* Patients with a personal or family history of inflammatory disease (SpA , ulcerative colitis , chron , PSO , RA, SAPHO)
* Patients with a history of trauma or surgery of the pelvis
* Pregnant women
* Women who gave birth over a year ago and less than 2 years ago

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 512 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Presence of MRI inflammatory and structural lesions of the sacroiliac joints (including pubic symphysis) in the population of women who gave birth within the past 12 months. | Time of MRI (within the year following childbirth or pregnancy)
  MRI Lesions will be analyzed according to ASAS criteria. Inflammatory lesions will be evaluated on STIR (or T2 fat sat or T2 dixon) sequences.
  Structural lesions will be evaluated on T1 weighted sequences

SECONDARY OUTCOMES:
Morphological analysis of sacroiliac lesions in women aged from 18-50 years old. | Time of MRI
  Morphological analysis will evaluate erosion, fat, condensation, bone marrow edema using a 3 point scale (0-mild-high) for their number or extension.
Topographical analysis of sacroiliac lesions in women aged from 18-50 years old. | Time of MRI
  Topographical analysis will assess the location : Iliac versus sacral, superior vs medial vs inferior, anterior vs posterior, pubic symphysis

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CYTEVAL, Principal Investigator — Montpellier University Hospital
Locations (1):
- Departement of Medical Imaging, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hoballah A, Lukas C, Leplat C, Taourel P, Pialat JB, Sans N, Ramos-Pascual S, Cyteval C. MRI of sacroiliac joints for the diagnosis of axial SpA: prevalence of inflammatory and structural lesions in nulliparous, early postpartum and late postpartum women. Ann Rheum Dis. 2020 Aug;79(8):1063-1069. doi: 10.1136/annrheumdis-2020-217208. Epub 2020 Jun 10. PMID 32522743